CLINICAL TRIAL: NCT03214211
Title: Assess the Long-term Safety and Efficacy of Pravafenix Cap. in Korean Patients With Dyslipidemia: a Multicenter, Prospective, Observational Study
Brief Title: Prospective Observational Study of Pravafenix Cap
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Yooyoung Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: YYPCT_APOLLO_OS
Record Dates: First submitted 2017-06-21; First posted 2017-07-11 (Actual); Last update posted 2017-08-31 (Actual); Status verified 2017-07

CONDITIONS: Dyslipidemias
MeSH Terms: conditions — Dyslipidemias

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To observe the effiacay, safety and risk of developing diabetes, review the patients chars who had administrated or neet to administrate the Pravafenix cap for enroll period, it is an prospective observational study that only collect the collectable information follwoing the hospital visiting date from enroll point to information collecting date. There is no extra visit for this study.

Observe the data which has been collected for 3 yearts every year from enroll point, if the patients agree to be participated in this study and are suitable in inclusion/exclusion criteria.

If the lipid-lowering drugs(only Ezetimibe is possible) is add-on the Pravafenix Cap administrating period, it will be analyzed by laering analysis separately. But, the reason why it is add-on to have to be written on e-CRF.

ELIGIBILITY:
Inclusion Criteria:

Among the patients with artheriosclerotic cardiovascular heart failure who have been hopitalized or visited the hospital.

1. Men or Women over 20 years old
2. Patients who had already administrated or need to administrate the Pravafenix Cap
3. Patients who have abnormal opinion(dyslipidemia) about LDL-C, TG, HDL-C at the enroll point

   * 70mg/dL ≤ LDL-C ≤ 160mg/dL
   * 150mg/dL ≤ TG ≤ 500mg/dL or HDL-C < 40mg/dL(Men), 50mg/dL(Women)
4. Voluntary written informed consent to study participation

Exclusion Criteria:

1. Patient who have hypersensitivity about Pravafenix Cap or ingredients of the Pravafenix Cap.
2. Patients suffer from liver disease (Biliary cirrhosis, activated hepatophay or lasting potentiation of the transaminase 3 times excess from normal valus(which has no cause).
3. Patients suffer from kidney disease(CCR < 60ml/min)
4. Patients have photo-allergy (allergic reaction causeed by sunlight or exposure to UV light) or phototoxic reactions (damage to skin caused by exposure to sunlight or UV light) during treatment with fibrates(lipid-modifying medicines) or ketoprofen (an anti-inflammatory medicine that can be used orally or on the skin for muscle and bone disorders, and orally for gout or period pain).
5. Acute or chronic patients who have high triglycerides academia.
6. Pregnant or breat-feeding
7. Someone who have a history of muscle problems during treatment with cholesterol-controlling medicines called 'statins' (such as simvastatin, atorvastatin, pravastatin or rosuvastatin) or fibrates (such as fenofibrate and bezafibrate).
8. Pateints who have uncontrolled hypothyroidism or hyperthyroidism.
9. Patinets who couldn't be participated in the study by the other opinion of the investigator.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have dyslipidemia, already administrated or need to administrate the Pravafenix Cap.
Sampling Method: Probability Sample
Enrollment: 3088 (Estimated)
Dates: Start 2017-08-30 (Estimated); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Occurrence and mortaity about the cardiovascular disease case for 3 years from administrating the Pravafenix Cap. | For 3 years
  (Occurence of the MACE for 3 years after aministrating the Pravfenix Cap)

SECONDARY OUTCOMES:
Variation of the diabetic index (Before/after the administration of the Pravafenix Cap) | For 3 years
  FBS, HbA1c
Variation of lipid parameter(Before/after the administration of the Pravafenix Cap) | For 3 years
  TC, LDL-C, TG, HDL-C
Variation of inflammatory index(Before/after the administration of the Pravafenix Cap) | For 3 years
  hs-CRP
Occurrence of the major clinical events | For 3 years
  eventsBefore/after the administration of the Pravafenix Cap.

CONTACTS AND LOCATIONS:
Overall Officials: Myung-Ho Jeong, Ph.D, Principal Investigator — Chonnam National University Hospital
Locations (1):
- Chonnam national university hospital, Gwangju, South Korea